CLINICAL TRIAL: NCT02927431
Title: A Phase II, Global, Randomized Study to Evaluate the Efficacy and Safety of Danirixin (GSK1325756) Co-administered With a Standard-of-care Antiviral (Oseltamivir), in the Treatment of Adults Hospitalized With Influenza
Brief Title: Study to Evaluate the Efficacy and Safety of Danirixin Co-administered With Oseltamivir in the Treatment of Adults Hospitalized With Influenza
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped early due to lack of enrollment.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201023; 2016-002512-40 (EudraCT Number)
Record Dates: First submitted 2016-09-29; First posted 2016-10-07 (Estimated); Results first posted 2018-07-02 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Virus Diseases
Keywords: Anti-inflammatory; Danirixin; Influenza; Hospitalized patients
MeSH Terms: conditions — Virus Diseases; Influenza, Human | interventions — danirixin; Oseltamivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Danirixin 15 mg FBE IV plus 75 mg oseltamivir (Experimental): Subjects will receive double blind 15 mg FBE IV danirixin twice daily with open label 75 mg oral oseltamivir twice daily for 5 days. If a subject is discharged from the hospital in less than 5 days, treatment with IV DNX will be discontinued.
  Interventions: Drug: Danirixin 15 mg FBE; Drug: Oseltamivir 75 mg
- Danirixin 50 mg FBE IV plus 75 mg oseltamivir (Experimental): Subjects will receive double blind 50 mg FBE IV danirixin twice daily with 75 mg oral oseltamivir twice daily for 5 days. If a subject is discharged from the hospital in less than 5 days, treatment with IV DNX will be discontinued.
  Interventions: Drug: Danirixin 50 mg FBE; Drug: Oseltamivir 75 mg
- Placebo of danirixin IV plus 75 mg oseltamivir (Placebo Comparator): Subjects will receive double blind IV placebo of DNX twice daily with 75 mg oral oseltamivir twice daily for 5 days. If a subject is discharged from the hospital in less than 5 days, treatment with IV DNX will be discontinued.
  Interventions: Drug: Placebo; Drug: Oseltamivir 75 mg

INTERVENTIONS:
Drug: Danirixin 15 mg FBE — This intervention is available as a 50 mg FBE sterile lyophilized powder containing DNX (hydrobromide salt hemihydrate) equivalent to 50mg of free base along with Beta-cyclodextrin sulfobutylether, mannitol, citric acid and sodium hydroxide. The formulation is supplied as lyophilized powder/cake contained in a 30mL vial. Each vial is reconstituted with 9.5 mL water for injection and further diluted with saline for IV infusion to provide a dose of 15 mg FBE.
  Arms: Danirixin 15 mg FBE IV plus 75 mg oseltamivir
Drug: Danirixin 50 mg FBE — This intervention is available as a 50 mg FBE sterile lyophilized powder containing DNX (hydrobromide salt hemihydrate) equivalent to 50mg of free base along with Beta-cyclodextrin sulfobutylether, mannitol, citric acid and sodium hydroxide. The formulation is supplied as lyophilized powder/cake contained in a 30mL vial. Each vial is reconstituted with 9.5 mL water for injection and further diluted with saline for IV infusion.
  Arms: Danirixin 50 mg FBE IV plus 75 mg oseltamivir
Drug: Placebo — No vials of placebo to match IV DNX will be provided. A normal saline solution of matched volume will be prepared by unblinded personnel at the site to act as a placebo to DNX. Clear solution of placebo will be administered as IV infusion.
  Arms: Placebo of danirixin IV plus 75 mg oseltamivir
Drug: Oseltamivir 75 mg — Oseltamivir (Tamiflu - manufactured by Roche) formulation is available as 75 mg Capsule and as powder for oral suspension. After constitution with 55 mL of water, each bottle delivers a usable volume of 60 mL of oral suspension equivalent to 360 mg oseltamivir base (6 mg/mL). No oseltamivir capsules or powder for oral suspension will be provided. Sites will source the OSV locally and it will be provided open-label.

SUMMARY:
Danirixin (DNX) is a novel, selective, and reversible antagonist of the C-X-C chemokine receptor (CXCR) 2 and has been shown to decrease neutrophil transmigration and activation to areas of inflammation. An intravenous (IV) formulation of DNX hydrobromide (HBr) is being developed as an anti-inflammatory agent for treatment of adults hospitalized with influenza (IFV). While early therapy with antivirals decreases severity and duration of symptoms of influenza, there are no drugs that have demonstrated clinical efficacy in randomized clinical trials in this population. Current treatment guidelines for hospitalized IFV recommend neuraminidase inhibitors as standard of care therapy. IFV studies in animals have demonstrated that therapeutic treatment with the combination of a CXCR2 antagonist and a neuraminidase inhibitor reduced lung neutrophils and showed trends for improvements in clinical scores, lung function and pathology with no evidence of worsening outcomes, including viral load. This Phase 2, randomized, double-blind (for IV DNX), placebo-controlled (for IV DNX) 3-arm study will be the first study to determine the efficacy and safety of IV DNX when co-administered (in all groups) with standard of care antiviral treatment (open-label oral oseltamivir [OSV]) in subjects hospitalized with IFV. The primary objective of the study is to assess the efficacy of treatment with IV DNX twice daily given with oral OSV compared to oral OSV twice daily on time to clinical response (TTCR). In this study, subjects will be randomized in a 2:2:1 ratio to 15 milligram (mg) free base equivalent (FBE) IV DNX, 50 mg FBE IV DNX, or matching placebo twice daily. All subjects will also receive open-label 75 mg oral OSV, twice daily (given as standard of care). The study treatment duration will be for up to 5 days. The investigator may elect to continue treatment with OSV after 5 days of study treatment. Follow up will continue until Day 45 for all subjects. The study will begin with enhanced safety monitoring in sentinel cohorts, leading to stepwise enrollment of subjects. Subjects will be enrolled based on increasing levels of renal impairment, and less severe hospitalized subjects will be enrolled prior to enrollment of critically ill subjects, as this is the first study conducted in the hospitalized population with severe IFV. Approximately 300 subjects are targeted to be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years (as per local laws) of age and older at the time of signing the informed consent.
* Presence of fever (>=38.0 degree Celsius [>=100.4 degree Fahrenheit] by any route) at Baseline (enrollment) or history of fever/feverishness during the 48 hours prior.
* Oxygen (O2) saturation <95% on room air by trans-cutaneous method OR need for any supplemental oxygenation (non-invasive ventilation, facemask, facetent, nasal canula, etc) or ventilator support (mechanical ventilation, bi-level positive airway pressure [BIPAP], continuous positive airway pressure [CPAP]) or increase in oxygen supplementation requirement of >=2 liters for subjects with chronic oxygen dependency. For those subjects with a history of chronic hypoxia (without supplemental oxygen), an oxygen saturation of at least 3% below the subject's historical baseline oxygen saturation.
* And at least 2 out of the following 3: respiratory rate >24 breaths per minute. For those subjects who require ventilator support or oxygen supplementation, this requirement is waived; heart rate >100 beats per minute; SBP <90 millimeters of mercury (mm Hg).
* Severity of symptoms at enrollment: 1) Less severe hospitalized subjects are those who (but not limited to): are hemodynamically stable; may require oxygenation with facemask, facetent, nasal canula, etc; may or may not have radiological signs of lower respiratory tract disease; or have exacerbation of underlying chronic disease, including asthma, chronic obstructive pulmonary disease (COPD), or other cardiovascular conditions not leading to hemodynamic compromise. 2) Critically ill hospitalized subjects are those who (but not limited to): require CPAP, BIPAP, mechanical ventilation; have hemodynamic instability (with or without pressor support); or have central nervous system involvement (example encephalopathy, encephalitis).
* Presence of influenza that in the Investigator's judgment requires hospitalization for treatment and supportive care
* Onset of influenza symptoms within 6 days prior to study enrolment. Symptoms may include cough, dyspnea, sore throat, feverishness, myalgias, headache, nasal symptoms (rhinorrhea, congestion), fatigue, diarrhea, nausea and vomiting.
* A positive result from a rapid influenza test (provided by GlaxoSmithKline [GSK]) or other available, local laboratory diagnostic test
* Baseline renal criteria as follows: 1) Sentinel Cohorts: Normal renal function: Baseline creatinine clearance within normal reference ranges (>=80 milliliter per minute (mL/min) for the first approximately 30 subjects enrolled; Mild renal impairment: Baseline creatinine clearance of 50-79 mL/min for the next approximately 10 subjects enrolled into the sentinel cohort; Moderate renal impairment: Baseline creatinine clearance of 30-49 mL/min for the next approximately 10 subjects enrolled into the sentinel cohort. 2) Post-sentinel cohorts: Normal renal function, mild or moderate renal impairment: creatinine clearance >30mL/min.
* Baseline Liver Function Tests: Subjects will be included if:

  1. ALT is <=5 times the upper limit of normal (ULN) and bilirubin is <=2 times the ULN
  2. ALT is >5 but <=8 times the ULN and bilirubin is < 1.5 times the ULN
* Male or Female subjects could be eligible if: Male subjects with female partners of child bearing potential must comply with the pre-specified highly effective contraception requirements from the time of first dose of study medication until at least 36 hours (five half-lives) after the last dose of study medication. 1) Vasectomy with documentation of azoospermia 2) Male condom plus partner use of one of the contraceptive options below: Contraceptive subdermal implant; Intrauterine device or intrauterine system; Oral Contraceptive, either combined or progestogen alone; Injectable progestogen; Contraceptive vaginal ring; Percutaneous contraceptive patches
* For females, non-reproductive potential defined as: 1) Pre-menopausal females with one of the following: Documented tubal ligation; Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion; Hysterectomy; Documented Bilateral Oophorectomy 2) Postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause (refer to laboratory reference ranges for confirmatory levels)]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. 3) Reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from the first dose of study medication until at least 36 hours after the last dose of study medication and completion of the post treatment (PT) Day 3 visit. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.
* Subjects willing and able to give written informed consent to participate in the study and to adhere to the procedures stated in the protocol OR Legally acceptable representative (LAR) willing and able to give written informed consent on behalf of the subject to participate in the study for unconscious adults, and those incapable of consenting themselves due to their medical condition (e.g. too weak or debilitated, severe shortness of breath), due to literacy issues or included as permitted by local regulatory authorities, institutional review board (IRB)/independent ethics committee (IECs) or local laws.
* French subjects: In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion Criteria:

* Subjects who, in the opinion of the investigator, are not likely to survive the next 48 hours beyond Baseline;
* Immunosuppression, whether due to primary immunosuppressive conditions, such as history of inherited immunodeficiency syndromes, human immunodeficiency virus (HIV) infection, or secondary conditions, such as immunosuppressive medication, stem cell or solid organ transplantation, or malignancy;
* Documented current liver disease (including Hepatitis A, B, or C), or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones);
* Baseline Liver Function Tests: Subjects will be excluded if:

  1. ALT >8 times the ULN
  2. Bilirubin is >2 times the ULN
* Corrected QT Interval (QTc) Criteria: Corrected QT Interval using Bazette's formula (QTcB) or Corrected QT Interval using Fridericia forumula (QTcF) >480 millisecond (msec) or >500 msec with bundle branch block;
* For subjects enrolled in the sentinel cohorts: diabetes mellitus and chronic kidney disease;
* Subjects who require dialysis, or are on renal replacement therapies;
* Subjects who require extra corporeal membrane oxygenation (ECMO) at baseline (enrolled subjects who subsequently require ECMO may continue in the study)
* Women who are pregnant as determined by a positive human chorionic gonadotrophin (hCG) ultrasensitive test prior to dosing or women who are breastfeeding;
* Subjects who received other treatments for influenza including vitaglutam, umifenovir, and neuraminidase inhibitors (oseltamivir, zanamivir, peramivir) for more than 72 hours during current acute illness;
* Subjects who received any immunoglobulins within 6 months of screening or planned administration of any of these products during the treatment period.
* Subjects treated with cytotoxic or immunosuppressive drugs within six months of study enrolment. Topical, intra-articularly injected, or inhaled glucocorticoids, topical calcineurin inhibitors or imiquimod are allowed.
* Known history of drug abuse within 6 months of study start.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Absolute neutrophil count <1.0 giga per Liter (Gi/L)
* Subjects who have participated in a clinical trial using an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2017-05-24 (Actual); Study Completion 2017-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- United States (5):
  - GSK Investigational Site, Stamford, Connecticut
  - GSK Investigational Site, Council Bluffs, Iowa
  - GSK Investigational Site, Natchitoches, Louisiana
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Salem, Virginia
- GSK Investigational Site, Bucharest, Romania
- GSK Investigational Site, Smolensk, Russia
- GSK Investigational Site, Lund, Sweden

REFERENCES:
- [Background] Madan A, Chen S, Yates P, Washburn ML, Roberts G, Peat AJ, Tao Y, Parry MF, Barnum O, McClain MT, Roy-Ghanta S. Efficacy and Safety of Danirixin (GSK1325756) Co-administered With Standard-of-Care Antiviral (Oseltamivir): A Phase 2b, Global, Randomized Study of Adults Hospitalized With Influenza. Open Forum Infect Dis. 2019 Apr 3;6(4):ofz163. doi: 10.1093/ofid/ofz163. eCollection 2019 Apr. PMID 31041358

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized study to evaluate the efficacy and safety of Danirixin (DNX) co-administered with a standard-of-care antiviral (oseltamivir [OSV]), in the treatment of adults hospitalized with influenza. The study enrolled participants in 7 centers across 3 countries (Romania,Sweden and United States) and was terminated due to poor enrollment
Pre-assignment Details: A total of 14 participants were screened for the study, of which 4 participants were screening failures. 10 participants received study treatment.
Groups:
- Placebo + OSV: Participants received matching placebo given as a 1 hour infusion twice daily for up to 5 days. Infusion was administered at a constant rate over approximately 1 hour +- 10 minutes and approximately 12 hours apart +- 1 hour. All participants also received open-label oral OSV 75 milligram (mg) twice daily given as standard of care. The investigator could elect to continue treatment with OSV after 5 days of study treatment.
- DNX 15 mg + OSV: Participants received DNX 15 mg given as a 1 hour infusion twice daily for up to 5 days. Infusion was administered at a constant rate over approximately 1 hour +- 10 minutes and approximately 12 hours apart +- 1 hour. All participants also received open-label oral OSV 75 mg twice daily given as standard of care. The investigator could elect to continue treatment with OSV after 5 days of study treatment.
- DNX 50 mg + OSV: Participants received DNX 50 mg given as a 1 hour infusion twice daily for up to 5 days. Infusion was administered at a constant rate over approximately 1 hour +- 10 minutes and approximately 12 hours apart +- 1 hour. All participants also received open-label oral OSV 75 mg twice daily given as standard of care. The investigator could elect to continue treatment with OSV after 5 days of study treatment.
Period: Overall Study
Arm/Group | Placebo + OSV | DNX 15 mg + OSV | DNX 50 mg + OSV
Started | 2 | 4 | 4
Completed | 2 | 4 | 3
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo + OSV: Participants received matching placebo given as a 1 hour infusion twice daily for up to 5 days. Infusion was administered at a constant rate over approximately 1 hour +- 10 minutes and approximately 12 hours apart +- 1 hour. All participants also received open-label oral OSV 75 mg twice daily given as standard of care. The investigator could elect to continue treatment with OSV after 5 days of study treatment.
- Total: Total of all reporting groups
Arm/Group | Placebo + OSV | DNX 15 mg + OSV | DNX 50 mg + OSV | Total
Number analyzed (Participants) | 2 | 4 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.0 (24.04) | 66.0 (8.76) | 63.0 (24.90) | 63.8 (17.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3 | 6
  Male | 1 | 2 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/ Ethnicity: African American/African Heritage | 1 | 0 | 1 | 2
  Race/ Ethnicity: Asian-Central/South Asian Heritage | 0 | 0 | 1 | 1
  Race/ Ethnicity: White-White/Caucasian/European Heritage | 1 | 4 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Time to Clinical Response (TTCR)
Description: The clinical response was defined as Hospital discharge due to clinical improvement OR normalization of temperature; and oxygen saturation; and respiratory status/heart rate/systolic blood pressure (normalization of 2 out of these 3 parameters). The clinical response based on vital signs/ventilation status required 24-hour confirmation. Considering 2-hour assessment window, the response confirmation period was 22 hours. Kaplan Meier estimates for the median of TTCR was provided. One participant had vital sign resolution at Baseline and was counted as having a clinical response but was not included in the Kaplan Meier Estimates. Influenza Positive Population (IPP) Population comprised of all participants in the Intent to Treat Exposed (ITT-E) Population with influenza infection (positive influenza Polymerase Chain Reaction [PCR] or culture at any time point) confirmed by central lab testing. Only those participants with data available at the indicated time point were analyzed.
Time Frame: Up to 45 Days
Population: IPP Population
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo + OSV | DNX 15 mg + OSV | DNX 50 mg + OSV
Number analyzed (Participants) | 2 | 3 | 4
Days | 1.33 [0.71 to 1.95] | 4.53 [2.95 to 5.71] | 4.76 [3.66 to 5.08]

2. Secondary Outcome: Time to Respiratory Response (TTRR)
Description: Time to Respiratory Response was defined as meeting at least one of the following criteria, and maintained for 24 hours: return to pre-morbid oxygen requirement (participants with chronic oxygen use or ventilator support), or return to no requirement of supplemental oxygen, or respiratory rate <=24 per minute (without supplemental oxygen). Kaplan Meier estimates for the median of TTRR for each treatment group was provided. NA indicates data is not available. Due to limited data, no TTRR estimate could be calculated for any of the treatment groups.
Time Frame: Up to 45 Days
Population: IPP Population
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Placebo + OSV | DNX 15 mg + OSV | DNX 50 mg + OSV
Number analyzed (Participants) | 2 | 4 | 4
Days | NA [1.95 to NA] — Data could not be calculated due to insufficient number of participants with events. | NA [1.07 to NA] — Data could not be calculated due to insufficient number of participants with events. | NA [3.04 to NA] — Data could not be calculated due to insufficient number of participants with events.

3. Secondary Outcome: Time to Absence of Fever
Description: Time from first dose of treatment to time to afebrile status (<=36.6 degree celsius-axilla/temporal or <=37.2 degree celsius- oral, or <=37.7 degree celsius-rectal/core, tympanic) was to be evaluated.
Time Frame: Up to 45 Days
Population: IPP Population. As the study was terminated, only a selected set of originally planned analysis were performed and hence this endpoint was not analyzed.
Arm/Group | Placebo + OSV | DNX 15 mg + OSV | DNX 50 mg + OSV
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Time to Improved Oxygen Saturation
Description: Time from first dose of treatment to time of improved oxygen saturation was to be calculated. A participant with a history of chronic hypoxia (without supplemental oxygen) satisfied normalization criteria for oxygen saturation if the value (without supplemental oxygen) is <=2 percent from participant's historical oxygen saturation Baseline as recorded within 12 months prior to enrollment as documented in the participant's medical records. This requirement was to be waived for participants with a history of chronic supplemental oxygen requirement who had a Baseline oxygen saturation <95 percent with supplemental oxygen, within 12 months prior to enrollment as documented in the participant's medical records.
Time Frame: Up to 45 Days
Population: as for outcome 3
Arm/Group | Placebo + OSV | DNX 15 mg + OSV | DNX 50 mg + OSV
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Time to Improved Heart Rate
Description: Time from first dose of treatment to time of heart rate <=100 beats per minute was to be evaluated.
Time Frame: Up to 45 Days
Population: as for outcome 3
Arm/Group | Placebo + OSV | DNX 15 mg + OSV | DNX 50 mg + OSV
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Time to Improved Systolic Blood Pressure (SBP)
Description: Time from first dose of treatment to time of SBP at >=90 millimeters of mercury (mmHg) was to be evaluated.
Time Frame: Up to 45 Days
Population: as for outcome 3
Arm/Group | Placebo + OSV | DNX 15 mg + OSV | DNX 50 mg + OSV
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Percentage of Participants With Clinical Response Over Time
Description: The clinical response was defined as Hospital discharge due to clinical improvement OR normalization of temperature; and oxygen saturation; and respiratory status/heart rate/systolic blood pressure (normalization of 2 out of these 3 parameters). The clinical response based on vital signs/ventilation status required 24-hour confirmation. Considering 2-hour assessment window, the response confirmation period was 22 hours. Percentage of participants with positive clinical response are presented.
Time Frame: Up to 45 Days
Population: IPP Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + OSV | DNX 15 mg + OSV | DNX 50 mg + OSV
Number analyzed (Participants) | 2 | 4 | 4
Percentage of Participants | 100 | 100 | 100

8. Secondary Outcome: Percentage of Participants With Improved Respiratory Status Over Time
Description: The Respiratory Response was defined as meeting at least one of the following criteria, and maintained for 24 hours: return to pre-morbid oxygen requirement (participants with chronic oxygen use or ventilator support), or return to no requirement of supplemental oxygen, or respiratory rate <=24 per minute (without supplemental oxygen). Percentage of participants with improved respiratory status has been presented.
Time Frame: Up to 45 Days
Population: IPP Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo + OSV | DNX 15 mg + OSV | DNX 50 mg + OSV
Number analyzed (Participants) | 2 | 4 | 4
Percentage of Participants | 50 | 50 | 50

9. Secondary Outcome: Time to Improvement of Ventilation Status
Description: Time to improvement of ventilation status was assessed by modality, frequencies and durations of invasive and non-invasive ventilator support, duration of oxygen supplementation.
Time Frame: Up to 45 Days
Population: as for outcome 3
Arm/Group | Placebo + OSV | DNX 15 mg + OSV | DNX 50 mg + OSV
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Number of Days of Stay in the Intensive Care Unit (ICU)
Description: Number of days of stay in the ICU over the treatment period and post treatment period was to be recorded.
Time Frame: Up to 45 Days
Population: as for outcome 3
Arm/Group | Placebo + OSV | DNX 15 mg + OSV | DNX 50 mg + OSV
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Number of Participants Requiring ICU Admission and Readmission
Description: Number of participants requiring ICU admission during treatment period and after post treatment was to be recorded.
Time Frame: Up to 45 Days
Population: as for outcome 3
Arm/Group | Placebo + OSV | DNX 15 mg + OSV | DNX 50 mg + OSV
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Number of Days of Stay in the Hospital
Description: Number of days of stay in the hospital over treatment period and post treatment period was to be recorded.
Time Frame: Up to 45 Days
Population: as for outcome 3
Arm/Group | Placebo + OSV | DNX 15 mg + OSV | DNX 50 mg + OSV
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Development of Septic Shock
Description: Development of septic shock was to be assessed by occurrence of hypotension requiring vasopressive therapy and serum lactate level >2 millimeter (mm) after adequate fluid resuscitation. Number of participants with development of septic shock were planned to be presented.
Time Frame: Up to 45 Days
Population: as for outcome 3
Arm/Group | Placebo + OSV | DNX 15 mg + OSV | DNX 50 mg + OSV
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Number of Participants Used Antibiotics for Complications of Influenza
Description: Complications of influenza such as bacterial pneumonia, pneumothorax, pleural effusion, acute respiratory distress syndrome (ARDS), myositis, encephalitis, myocarditis, and associated antibiotic use was recorded. Number of participants who reqruied use of associated antibiotics for complications of influenza is presented.
Time Frame: Up to 45 Days
Population: IPP Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + OSV | DNX 15 mg + OSV | DNX 50 mg + OSV
Number analyzed (Participants) | 2 | 4 | 4
Participants | 1 | 1 | 1

15. Secondary Outcome: Number of Participants With Improvement in Ordinal Scale of Clinical Efficacy Over Time
Description: Number of participants with improvement in ordinal scale of clinical efficacy over time was to be assessed by: death, mechanical vent, in the ICU, non-ICU hospitalization, and hospital discharge.
Time Frame: Up to 45 Days
Population: as for outcome 3
Arm/Group | Placebo + OSV | DNX 15 mg + OSV | DNX 50 mg + OSV
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Any Non-serious Adverse Event (AE); Any Serious AE (SAE); Any AEs of Special Interest (AESIs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, any other situation according to medical or scientific judgment that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention or event associated with liver injury and impaired liver function were categorized as SAE. Participants who received any of the study treatment and had any AE or SAE or AESI were considered for analysis. Safety Population comprised of all participants who received at least 1 dose of study treatment.
Time Frame: Up to 45 Days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + OSV | DNX 15 mg + OSV | DNX 50 mg + OSV
Number analyzed (Participants) | 2 | 4 | 4
Participants
  Any non-SAE | 0 | 4 | 4
  Any SAE | 0 | 0 | 2
  Any AESI | 0 | 1 | 1

17. Secondary Outcome: Change From Baseline in Albumin and Total Protein
Description: Blood samples were collected to evaluate albumin and total protein at indicated time points. Values at Day 1 were considered as Baseline values. Change from Baseline at each visit was calculated by subtracting Baseline value from post-dose visit value. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates data is not available.
Time Frame: Baseline and up to 45 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Gram per Liter (G/L)
Arm/Group | Placebo + OSV | DNX 15 mg + OSV | DNX 50 mg + OSV
Number analyzed (Participants) | 2 | 4 | 4
Gram per Liter (G/L)
  Albumin, Day 2, n=1,0,0: number analyzed (Participants) | 1 | 0 | 0
  Albumin, Day 2, n=1,0,0 | 2.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. |  |
  Albumin, Day 2, sample 2, n=0,0,1: number analyzed (Participants) | 0 | 0 | 1
  Albumin, Day 2, sample 2, n=0,0,1 |  |  | 0.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated.
  Albumin, Day 3, n=1,2,2: number analyzed (Participants) | 1 | 2 | 2
  Albumin, Day 3, n=1,2,2 | 0.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -5.0 (1.41) | -2.0 (2.83)
  Albumin, Day 3, sample 2, n=0,1,2: number analyzed (Participants) | 0 | 1 | 2
  Albumin, Day 3, sample 2, n=0,1,2 |  | -9.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -4.5 (4.95)
  Albumin, Day 4, n=0,1,2: number analyzed (Participants) | 0 | 1 | 2
  Albumin, Day 4, n=0,1,2 |  | -1.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -3.0 (4.24)
  Albumin, Day 4, sample 2, n=0,1,1: number analyzed (Participants) | 0 | 1 | 1
  Albumin, Day 4, sample 2, n=0,1,1 |  | -8.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -5.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated.
  Albumin, Day 5, n=1,1,3: number analyzed (Participants) | 1 | 1 | 3
  Albumin, Day 5, n=1,1,3 | 0.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -5.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -3.7 (6.03)
  Albumin, Day 6, n=1,1,4: number analyzed (Participants) | 1 | 1 | 4
  Albumin, Day 6, n=1,1,4 | 1.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -6.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -2.8 (4.99)
  Albumin, Day 7, n=1,1,1: number analyzed (Participants) | 1 | 1 | 1
  Albumin, Day 7, n=1,1,1 | -2.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -5.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -3.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated.
  Albumin, Day 8, n=1,0,0: number analyzed (Participants) | 1 | 0 | 0
  Albumin, Day 8, n=1,0,0 | 0.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. |  |
  Albumin, Discharge/Day 45, n=2,2,3: number analyzed (Participants) | 2 | 2 | 3
  Albumin, Discharge/Day 45, n=2,2,3 | 2.5 (2.12) | -0.5 (0.71) | 5.7 (6.81)
  Albumin, Day 3 post last dose, n=1,3,3: number analyzed (Participants) | 1 | 3 | 3
  Albumin, Day 3 post last dose, n=1,3,3 | 0.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -1.3 (1.15) | -2.3 (1.15)
  Total Protein, Day 2, n=1,0,1: number analyzed (Participants) | 1 | 0 | 1
  Total Protein, Day 2, n=1,0,1 | 1.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. |  | -1.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated.
  Total Protein, Day 3, n=1,2,2: number analyzed (Participants) | 1 | 2 | 2
  Total Protein, Day 3, n=1,2,2 | 1.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -5.5 (4.95) | -3.0 (4.24)
  Total Protein, Day 3, sample 2, n=0,1,2: number analyzed (Participants) | 0 | 1 | 2
  Total Protein, Day 3, sample 2, n=0,1,2 |  | -13.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -4.0 (4.24)
  Total Protein, Day 4, n=0,1,2: number analyzed (Participants) | 0 | 1 | 2
  Total Protein, Day 4, n=0,1,2 |  | -1.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -4.0 (5.66)
  Total Protein, Day 4, sample 2, n=0,1,1: number analyzed (Participants) | 0 | 1 | 1
  Total Protein, Day 4, sample 2, n=0,1,1 |  | -10.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -7.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated.
  Total Protein, Day 5, n=1,1,3: number analyzed (Participants) | 1 | 1 | 3
  Total Protein, Day 5, n=1,1,3 | -1.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -7.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -5.7 (10.97)
  Total Protein, Day 6, n=1,1,4: number analyzed (Participants) | 1 | 1 | 4
  Total Protein, Day 6, n=1,1,4 | 0.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -7.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -4.0 (6.98)
  Total Protein, Day 7, n=1,1,1: number analyzed (Participants) | 1 | 1 | 1
  Total Protein, Day 7, n=1,1,1 | -3.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -5.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -2.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated.
  Total Protein, Day 8, n=1,0,0: number analyzed (Participants) | 1 | 0 | 0
  Total Protein, Day 8, n=1,0,0 | 0.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. |  |
  Total Protein, Discharge/Day 45, n=2,2,3: number analyzed (Participants) | 2 | 2 | 3
  Total Protein, Discharge/Day 45, n=2,2,3 | 0.0 (2.83) | -1.5 (2.12) | 6.7 (11.02)
  Total Protein, Day 3 post last dose, n=1,3,3: number analyzed (Participants) | 1 | 3 | 3
  Total Protein, Day 3 post last dose, n=1,3,3 | -0.3 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -3.0 (2.00) | -3.3 (3.51)

18. Secondary Outcome: Change From Baseline in White Blood Cell Count (WBC) and Absolute Neutrophil Count (ANC)
Description: Blood samples were collected to evaluate WBC and ANC at indicated time points. Values at Day 1 were considered as Baseline values. Change from Baseline at each visit was calculated by subtracting Baseline value from post-dose visit value. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates data is not available.
Time Frame: Baseline and up to 45 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Giga cells per Liter (GI/L)
Arm/Group | Placebo + OSV | DNX 15 mg + OSV | DNX 50 mg + OSV
Number analyzed (Participants) | 2 | 4 | 4
Giga cells per Liter (GI/L)
  WBC, Day 2, n=1,0,0: number analyzed (Participants) | 1 | 0 | 0
  WBC, Day 2, n=1,0,0 | -2.70 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. |  |
  WBC, Day 3, n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  WBC, Day 3, n=1,1,0 | -5.10 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -3.00 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. |
  WBC, Day 4, n=0,2,1: number analyzed (Participants) | 0 | 2 | 1
  WBC, Day 4, n=0,2,1 |  | 1.15 (3.889) | -7.10 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated.
  WBC, Day 5, n=1,1,1: number analyzed (Participants) | 1 | 1 | 1
  WBC, Day 5, n=1,1,1 | -2.90 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -3.70 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -5.30 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated.
  WBC, Day 6, n=1,0,0: number analyzed (Participants) | 1 | 0 | 0
  WBC, Day 6, n=1,0,0 | -2.40 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. |  |
  WBC, Day 7, n=1,0,0: number analyzed (Participants) | 1 | 0 | 0
  WBC, Day 7, n=1,0,0 | -2.90 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. |  |
  WBC, Day 8, n=1,0,0: number analyzed (Participants) | 1 | 0 | 0
  WBC, Day 8, n=1,0,0 | -3.10 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. |  |
  WBC, Discharge/Day 45, n=2,3,1: number analyzed (Participants) | 2 | 3 | 1
  WBC, Discharge/Day 45, n=2,3,1 | -3.55 (2.051) | 3.97 (2.765) | -9.50 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated.
  WBC, Day 3 post last dose, n=1,4,1: number analyzed (Participants) | 1 | 4 | 1
  WBC, Day 3 post last dose, n=1,4,1 | -4.60 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | 1.95 (2.594) | -8.00 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated.
  ANC, Day 2, n=1,0,0: number analyzed (Participants) | 1 | 0 | 0
  ANC, Day 2, n=1,0,0 | -3.880 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. |  |
  ANC, Day 3, n=1,1,0: number analyzed (Participants) | 1 | 1 | 0
  ANC, Day 3, n=1,1,0 | -5.640 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -4.070 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. |
  ANC, Day 4, n=0,2,1: number analyzed (Participants) | 0 | 2 | 1
  ANC, Day 4, n=0,2,1 |  | 1.410 (3.2810) | -7.420 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated.
  ANC, Day 5, n=1,1,1: number analyzed (Participants) | 1 | 1 | 1
  ANC, Day 5, n=1,1,1 | -4.250 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -4.250 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -6.260 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated.
  ANC, Day 6, n=1,0,0: number analyzed (Participants) | 1 | 0 | 0
  ANC, Day 6, n=1,0,0 | -3.540 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. |  |
  ANC, Day 7, n=1,0,0: number analyzed (Participants) | 1 | 0 | 0
  ANC, Day 7, n=1,0,0 | -4.180 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. |  |
  ANC, Day 8, n=1,0,0: number analyzed (Participants) | 1 | 0 | 0
  ANC, Day 8, n=1,0,0 | -4.580 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. |  |
  ANC, Discharge/Day 45, n=2,3,1: number analyzed (Participants) | 2 | 3 | 1
  ANC, Discharge/Day 45, n=2,3,1 | -4.650 (1.9092) | 3.050 (2.9511) | -9.720 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated.
  ANC, Day 3 post last dose, n=1,4,1: number analyzed (Participants) | 1 | 4 | 1
  ANC, Day 3 post last dose, n=1,4,1 | -5.680 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | 1.033 (2.9818) | -9.060 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated.

19. Secondary Outcome: Change From Baseline in Total Bilirubin (T. Bilirubin), Creatinine and Direct Bilirubin (D. Bilirubin)
Description: Blood samples were collected to evaluate T. Bilirubin, creatinine and D. Bilirubin at indicated time points. Values at Day 1 were considered as Baseline values. Change from Baseline at each visit was calculated by subtracting Baseline value from post-dose visit value. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates data is not available.
Time Frame: Baseline and up to 45 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Micromole per Liter (µmol/L)
Arm/Group | Placebo + OSV | DNX 15 mg + OSV | DNX 50 mg + OSV
Number analyzed (Participants) | 2 | 4 | 4
Micromole per Liter (µmol/L)
  D. Bilirubin, Day 2, n=1,0,0: number analyzed (Participants) | 1 | 0 | 0
  D. Bilirubin, Day 2, n=1,0,0 | -2.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. |  |
  D. Bilirubin, Day 2, sample 2, n=0,0,1: number analyzed (Participants) | 0 | 0 | 1
  D. Bilirubin, Day 2, sample 2, n=0,0,1 |  |  | 0.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated.
  D. Bilirubin, Day 3, n=1,2,2: number analyzed (Participants) | 1 | 2 | 2
  D. Bilirubin, Day 3, n=1,2,2 | -2.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -2.0 (0.00) | 0.0 (2.83)
  D. Bilirubin, Day 3, sample 2, n=0,1,2: number analyzed (Participants) | 0 | 1 | 2
  D. Bilirubin, Day 3, sample 2, n=0,1,2 |  | -2.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | 0.0 (2.83)
  D. Bilirubin, Day 4, n=0,1,2: number analyzed (Participants) | 0 | 1 | 2
  D. Bilirubin, Day 4, n=0,1,2 |  | 0.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | 0.0 (0.00)
  D. Bilirubin, Day 4, sample 2, n=0,1,1: number analyzed (Participants) | 0 | 1 | 1
  D. Bilirubin, Day 4, sample 2, n=0,1,1 |  | -2.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -2.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated.
  D. Bilirubin, Day 5, n=1,1,3: number analyzed (Participants) | 1 | 1 | 3
  D. Bilirubin, Day 5, n=1,1,3 | 0.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | 0.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | 0.0 (2.00)
  D. Bilirubin, Day 6, n=1,1,4: number analyzed (Participants) | 1 | 1 | 4
  D. Bilirubin, Day 6, n=1,1,4 | 0.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | 0.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -0.5 (1.91)
  D. Bilirubin, Day 7, n=1,1,1: number analyzed (Participants) | 1 | 1 | 1
  D. Bilirubin, Day 7, n=1,1,1 | 0.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | 0.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | 2.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated.
  D. Bilirubin, Day 8, n=1,0,0: number analyzed (Participants) | 1 | 0 | 0
  D. Bilirubin, Day 8, n=1,0,0 | -2.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. |  |
  D. Bilirubin, Discharge/Day 45, n=2,2,3: number analyzed (Participants) | 2 | 2 | 3
  D. Bilirubin, Discharge/Day 45, n=2,2,3 | -3.0 (4.24) | -1.0 (1.41) | -0.7 (1.15)
  D. Bilirubin, Day 3 post last dose, n=1,3,3: number analyzed (Participants) | 1 | 3 | 3
  D. Bilirubin, Day 3 post last dose, n=1,3,3 | 0.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | 0.0 (0.00) | 0.7 (2.31)
  T. Bilirubin, Day 2, n=1,0,0: number analyzed (Participants) | 1 | 0 | 0
  T. Bilirubin, Day 2, n=1,0,0 | 0.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. |  |
  T. Bilirubin, Day 2, sample 2, n=0,0,1: number analyzed (Participants) | 0 | 0 | 1
  T. Bilirubin, Day 2, sample 2, n=0,0,1 |  |  | -4.00 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated.
  T. Bilirubin, Day 3, n=1,2,2: number analyzed (Participants) | 1 | 2 | 2
  T. Bilirubin, Day 3, n=1,2,2 | -2.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -2.0 (2.828) | -1.00 (1.414)
  T. Bilirubin, Day 3, sample 2, n=0,1,2: number analyzed (Participants) | 0 | 1 | 2
  T. Bilirubin, Day 3, sample 2, n=0,1,2 |  | -6.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -2.00 (0.000)
  T. Bilirubin, Day 4, n=0,1,2: number analyzed (Participants) | 0 | 1 | 2
  T. Bilirubin, Day 4, n=0,1,2 |  | 0.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -2.00 (2.828)
  T. Bilirubin, Day 4, sample 2, n=0,1,1: number analyzed (Participants) | 0 | 1 | 1
  T. Bilirubin, Day 4, sample 2, n=0,1,1 |  | -6.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | 0.00 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated.
  T. Bilirubin, Day 5, n=1,1,3: number analyzed (Participants) | 1 | 1 | 3
  T. Bilirubin, Day 5, n=1,1,3 | 0.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -2.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | 0.67 (1.155)
  T. Bilirubin, Day 6, n=1,1,4: number analyzed (Participants) | 1 | 1 | 4
  T. Bilirubin, Day 6, n=1,1,4 | -2.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | 2.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -0.50 (1.000)
  T. Bilirubin, Day 7, n=1,1,1: number analyzed (Participants) | 1 | 1 | 1
  T. Bilirubin, Day 7, n=1,1,1 | -6.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | 2.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | 0.00 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated.
  T. Bilirubin, Day 8, n=1,0,0: number analyzed (Participants) | 1 | 0 | 0
  T. Bilirubin, Day 8, n=1,0,0 | -6.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. |  |
  T. Bilirubin, Discharge/Day 45, n=2,2,3: number analyzed (Participants) | 2 | 2 | 3
  T. Bilirubin, Discharge/Day 45, n=2,2,3 | -1.0 (1.414) | 0.0 (2.828) | -0.67 (1.155)
  T. Bilirubin, Day 3 post last dose, n=1,3,3: number analyzed (Participants) | 1 | 3 | 3
  T. Bilirubin, Day 3 post last dose, n=1,3,3 | -4.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | 0.0 (2.000) | -4.60 (4.503)
  Creatinine, Day 2, n=2,2,4: number analyzed (Participants) | 2 | 2 | 4
  Creatinine, Day 2, n=2,2,4 | -7.95 (18.738) | -0.50 (5.657) | -3.35 (1.323)
  Creatinine, Day 2, sample 2, n=1,1,2: number analyzed (Participants) | 1 | 1 | 2
  Creatinine, Day 2, sample 2, n=1,1,2 | 3.50 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | 7.90 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -8.40 (0.566)
  Creatinine, Day 3, n=1,2,3: number analyzed (Participants) | 1 | 2 | 3
  Creatinine, Day 3, n=1,2,3 | -33.60 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -3.60 (1.273) | -4.77 (1.012)
  Creatinine, Day 3, sample 2, n=0,2,4: number analyzed (Participants) | 0 | 2 | 4
  Creatinine, Day 3, sample 2, n=0,2,4 |  | -9.30 (6.930) | 1.32 (8.397)
  Creatinine, Day 4, n=1,3,4: number analyzed (Participants) | 1 | 3 | 4
  Creatinine, Day 4, n=1,3,4 | -39.80 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -5.90 (6.222) | -4.20 (6.975)
  Creatinine, Day 4, sample 2, n=0,2,3: number analyzed (Participants) | 0 | 2 | 3
  Creatinine, Day 4, sample 2, n=0,2,3 |  | 0.45 (15.627) | -2.40 (7.375)
  Creatinine, Day 5, n=1,2,3: number analyzed (Participants) | 1 | 2 | 3
  Creatinine, Day 5, n=1,2,3 | -40.60 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -1.35 (9.405) | -2.67 (4.070)
  Creatinine, Day 5, sample 2, n=0,1,0: number analyzed (Participants) | 0 | 1 | 0
  Creatinine, Day 5, sample 2, n=0,1,0 |  | -15.90 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. |
  Creatinine, Day 6, n=1,1,4: number analyzed (Participants) | 1 | 1 | 4
  Creatinine, Day 6, n=1,1,4 | -44.20 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -10.60 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | 3.52 (4.396)
  Creatinine, Day 7, n=1,1,1: number analyzed (Participants) | 1 | 1 | 1
  Creatinine, Day 7, n=1,1,1 | -38.00 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -10.60 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -1.80 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated.
  Creatinine, Day 8, n=1,0,0: number analyzed (Participants) | 1 | 0 | 0
  Creatinine, Day 8, n=1,0,0 | -26.50 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. |  |
  Creatinine, Discharge/Day 45, n=2,2,3: number analyzed (Participants) | 2 | 2 | 3
  Creatinine, Discharge/Day 45, n=2,2,3 | -16.80 (22.486) | -3.55 (8.697) | 6.50 (4.521)
  Creatinine, Day 3 post last dose, n=1,3,3: number analyzed (Participants) | 1 | 3 | 3
  Creatinine, Day 3 post last dose, n=1,3,3 | -23.00 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -4.47 (9.750) | 2.93 (9.304)

20. Secondary Outcome: Change From Baseline in Alanine Amino Transferase (ALT), Aspartate Amino Transferase (AST) and Alkaline Phosphatase (ALP)
Description: Blood samples were collected to evaluate ALT, AST and ALP at indicated time points. Values at Day 1 were considered as Baseline values. Change from Baseline at each visit was calculated by subtracting Baseline value from post-dose visit value. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles). NA indicates data is not available.
Time Frame: Baseline and up to 45 days
Population: Safety Population
Measure: Mean (Standard Deviation); unit: International unit per Liter (IU/L)
Arm/Group | Placebo + OSV | DNX 15 mg + OSV | DNX 50 mg + OSV
Number analyzed (Participants) | 2 | 4 | 4
International unit per Liter (IU/L)
  ALT, Day 2, n=1,0,0: number analyzed (Participants) | 1 | 0 | 0
  ALT, Day 2, n=1,0,0 | 10.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. |  |
  ALT, Day 2, sample 2, n=0,0,1: number analyzed (Participants) | 0 | 0 | 1
  ALT, Day 2, sample 2, n=0,0,1 |  |  | -1.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated.
  ALT, Day 3, n=1,2,2: number analyzed (Participants) | 1 | 2 | 2
  ALT, Day 3, n=1,2,2 | 4.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | 3.0 (1.41) | 2.0 (5.66)
  ALT, Day 3, sample 2, n=0,1,2: number analyzed (Participants) | 0 | 1 | 2
  ALT, Day 3, sample 2, n=0,1,2 |  | -1.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -1.0 (5.66)
  ALT, Day 4, n=0,1,2: number analyzed (Participants) | 0 | 1 | 2
  ALT, Day 4, n=0,1,2 |  | -18.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -3.5 (2.12)
  ALT, Day 4, sample 2, n=0,1,1: number analyzed (Participants) | 0 | 1 | 1
  ALT, Day 4, sample 2, n=0,1,1 |  | 1.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | 10.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated.
  ALT, Day 5, n=1,1,3: number analyzed (Participants) | 1 | 1 | 3
  ALT, Day 5, n=1,1,3 | 0.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -2.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -0.3 (3.79)
  ALT, Day 6, n=1,1,4: number analyzed (Participants) | 1 | 1 | 4
  ALT, Day 6, n=1,1,4 | -1.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -37.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -2.3 (3.86)
  ALT, Day 7, n=1,1,1: number analyzed (Participants) | 1 | 1 | 1
  ALT, Day 7, n=1,1,1 | -2.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -42.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -6.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated.
  ALT, Day 8, n=1,0,0: number analyzed (Participants) | 1 | 0 | 0
  ALT, Day 8, n=1,0,0 | -1.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. |  |
  ALT, Discharge/Day 45, n=2,2,3: number analyzed (Participants) | 2 | 2 | 3
  ALT, Discharge/Day 45, n=2,2,3 | -6.0 (4.24) | -30.0 (35.36) | 0.7 (2.08)
  ALT, Day 3 post last dose, n=1,3,3: number analyzed (Participants) | 1 | 3 | 3
  ALT, Day 3 post last dose, n=1,3,3 | 2.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -17.0 (19.08) | -4.0 (3.61)
  AST, Day 2, n=1,0,0: number analyzed (Participants) | 1 | 0 | 0
  AST, Day 2, n=1,0,0 | 14.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. |  |
  AST, Day 2, sample 2, n=0,0,1: number analyzed (Participants) | 0 | 0 | 1
  AST, Day 2, sample 2, n=0,0,1 |  |  | -4.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated.
  AST, Day 3, n=1,2,2: number analyzed (Participants) | 1 | 2 | 2
  AST, Day 3, n=1,2,2 | 11.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | 6.0 (8.49) | -2.0 (2.83)
  AST, Day 3, sample 2, n=0,1,2: number analyzed (Participants) | 0 | 1 | 2
  AST, Day 3, sample 2, n=0,1,2 |  | 8.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -1.5 (4.95)
  AST, Day 4, n=0,1,2: number analyzed (Participants) | 0 | 1 | 2
  AST, Day 4, n=0,1,2 |  | -29.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -8.0 (2.83)
  AST, Day 4, sample 2, n=0,1,1: number analyzed (Participants) | 0 | 1 | 1
  AST, Day 4, sample 2, n=0,1,1 |  | 16.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | 0.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated.
  AST, Day 5, n=1,1,3: number analyzed (Participants) | 1 | 1 | 3
  AST, Day 5, n=1,1,3 | -10.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -9.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -7.3 (2.08)
  AST, Day 6, n=1,1,4: number analyzed (Participants) | 1 | 1 | 4
  AST, Day 6, n=1,1,4 | -12.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -46.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -5.8 (7.32)
  AST, Day 7, n=1,1,1: number analyzed (Participants) | 1 | 1 | 1
  AST, Day 7, n=1,1,1 | -11.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -51.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -11.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated.
  AST, Day 8, n=1,0,0: number analyzed (Participants) | 1 | 0 | 0
  AST, Day 8, n=1,0,0 | -12.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. |  |
  AST, Discharge/Day 45, n=2,2,3: number analyzed (Participants) | 2 | 2 | 3
  AST, Discharge/Day 45, n=2,2,3 | -12.0 (11.31) | -27.5 (30.41) | -3.0 (5.57)
  AST, Day 3 post last dose, n=1,3,3: number analyzed (Participants) | 1 | 3 | 3
  AST, Day 3 post last dose, n=1,3,3 | -10.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -21.7 (23.76) | -10.7 (5.86)
  ALP, Day 2, n=1,0,0: number analyzed (Participants) | 1 | 0 | 0
  ALP, Day 2, n=1,0,0 | 8.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. |  |
  ALP, Day 2,sample 2, n=0,0,1: number analyzed (Participants) | 0 | 0 | 1
  ALP, Day 2,sample 2, n=0,0,1 |  |  | -3.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated.
  ALP, Day 3, n=1,2,2: number analyzed (Participants) | 1 | 2 | 2
  ALP, Day 3, n=1,2,2 | 2.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -6.0 (8.49) | -8.0 (2.83)
  ALP, Day 3, sample 2, n=0,1,2: number analyzed (Participants) | 0 | 1 | 2
  ALP, Day 3, sample 2, n=0,1,2 |  | -23.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -14.0 (7.07)
  ALP, Day 4, n=0,1,2: number analyzed (Participants) | 0 | 1 | 2
  ALP, Day 4, n=0,1,2 |  | -25.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -5.5 (0.71)
  ALP, Day 4, sample 2, n=0,1,1: number analyzed (Participants) | 0 | 1 | 1
  ALP, Day 4, sample 2, n=0,1,1 |  | -22.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -4.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated.
  ALP, Day 5, n=1,1,3: number analyzed (Participants) | 1 | 1 | 3
  ALP, Day 5, n=1,1,3 | 6.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -8.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -11.0 (7.81)
  ALP, Day 6, n=1,1,4: number analyzed (Participants) | 1 | 1 | 4
  ALP, Day 6, n=1,1,4 | 5.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -51.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -9.5 (8.19)
  ALP, Day 7, n=1,1,1: number analyzed (Participants) | 1 | 1 | 1
  ALP, Day 7, n=1,1,1 | 2.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -50.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | 17.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated.
  ALP, Day 8, n=1,0,0: number analyzed (Participants) | 1 | 0 | 0
  ALP, Day 8, n=1,0,0 | 3.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. |  |
  ALP, Discharge/Day 45, n=2,2,3: number analyzed (Participants) | 2 | 2 | 3
  ALP, Discharge/Day 45, n=2,2,3 | 10.0 (0.00) | -25.5 (30.41) | 2.0 (9.64)
  ALP, Day 3 post last dose, n=1,3,3: number analyzed (Participants) | 1 | 3 | 3
  ALP, Day 3 post last dose, n=1,3,3 | 1.0 (NA) — NA indicates that data were not available as n=1 at this timepoint and standard deviation could not be calculated. | -19.7 (22.03) | -9.3 (7.51)

21. Secondary Outcome: Number of Participants With Clinically Significant Abnormality in Electrocardiogram (ECG)
Description: Single 12-lead ECGs were obtained at Baseline and on the day of last dose during the study using an ECG machine that automatically calculates the heart rate (HR) and measures PR, QRS, QT, and QT duration corrected for heart rate (QTc). Number of participants with clinically significant abnormality in ECG are presented.
Time Frame: Up to 6 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + OSV | DNX 15 mg + OSV | DNX 50 mg + OSV
Number analyzed (Participants) | 2 | 4 | 4
Participants | 0 | 0 | 1

22. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Intravenous (IV) DNX
Description: Cmax of IV DNX was to be derived from the Pharmacokinetics (PK) samples collected at Day 1 pre-dose, Day 3 at pre-dose and 0.5, 1, 1.5, 2, 3, 4, 8 and 12 hours post-dose and Day 5 pre-dose. PK Population comprised of all participants who underwent blood PK sampling during the study and from whom one or more blood concentration was determined.
Time Frame: Day 1 pre-dose, Day 3 at pre-dose and 0.5, 1, 1.5, 2, 3, 4, 8 and 12 hours post-dose and Day 5 pre-dose
Population: PK Population. As the study was terminated, only a selected set of originally planned analysis were performed and hence this endpoint was not analyzed due to limited sample size.
Arm/Group | DNX 15 mg + OSV | DNX 50 mg + OSV
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Area Under the Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC [0-t]) of IV DNX
Description: AUC (0-t) of IV DNX was to be derived from the PK samples collected at Day 1 pre-dose, Day 3 at pre-dose and 0.5, 1, 1.5, 2, 3, 4, 8 and 12 hours post-dose and Day 5 pre-dose.
Time Frame: Day 1 pre-dose, Day 3 at pre-dose and 0.5, 1, 1.5, 2, 3, 4, 8 and 12 hours post-dose and Day 5 pre-dose
Population: as for outcome 22
Arm/Group | DNX 15 mg + OSV | DNX 50 mg + OSV
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Time to Reach Cmax (Tmax) of IV DNX
Description: Tmax of IV DNX was to be derived from the PK samples collected at Day 1 pre-dose, Day 3 at pre-dose and 0.5, 1, 1.5, 2, 3, 4, 8 and 12 hours post-dose and Day 5 pre-dose.
Time Frame: Day 1 pre-dose, Day 3 at pre-dose and 0.5, 1, 1.5, 2, 3, 4, 8 and 12 hours post-dose and Day 5 pre-dose
Population: PK Population. As the study was terminated, only a selected set of originally planned analysis were performed and hence this endpoint was not analyzed due to limited PK parameters available.
Arm/Group | DNX 15 mg + OSV | DNX 50 mg + OSV
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Average Concentration (Cavg) of IV DNX
Description: Cavg of IV DNX was to be derived from the PK samples collected at Day 1 pre-dose, Day 3 at pre-dose and 0.5, 1, 1.5, 2, 3, 4, 8 and 12 hours post-dose and Day 5 pre-dose.
Time Frame: Day 1 pre-dose, Day 3 at pre-dose and 0.5, 1, 1.5, 2, 3, 4, 8 and 12 hours post-dose and Day 5 pre-dose
Population: as for outcome 22
Arm/Group | DNX 15 mg + OSV | DNX 50 mg + OSV
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: On-treatment SAEs and non-serious AEs were collected from the start of the study treatment up to Day 45.
Description: On treatment SAEs and non-serious AEs were reported for the Safety Population.
Arm/Group | Placebo + OSV | DNX 15 mg + OSV | DNX 50 mg + OSV
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/4 | 2/4
Other Adverse Events (participants affected / at risk) | 0/2 | 4/4 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + OSV (N=2) | DNX 15 mg + OSV (N=4) | DNX 50 mg + OSV (N=4)
Cardiac failure (Cardiac disorders) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + OSV (N=2) | DNX 15 mg + OSV (N=4) | DNX 50 mg + OSV (N=4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 1
Infusion site extravasation (General disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Monocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Interpretation of data is limited by the few participants enrolled prior to termination of the study due to poor recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-07-12): https://cdn.clinicaltrials.gov/large-docs/31/NCT02927431/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT02927431/SAP_001.pdf